CLINICAL TRIAL: NCT04141891
Title: Decision Making Among Older Adults: the AUTO Study
Brief Title: Advancing Understanding of Transportation Options
Acronym: AUTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19-0059; R01AG059613 (NIH)
Record Dates: First submitted 2019-10-22; First posted 2019-10-28 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Retinopathy; Macular Degeneration; Glaucoma; Retinitis Pigmentosa; Vision Disorders; Acute Coronary Syndrome; Implantable Defibrillator User; Congestive Heart Failure; Hypertrophic Obstructive Cardiomyopathy; Orthostatic Hypotension; Syncope; Presyncope; Narcolepsy; Dementia; Multiple Sclerosis; Parkinson Disease; Brain Injuries; Spinal Cord Injuries; Stroke; Vertigo; Dizziness; Seizures; Substance Use; Insulin Dependent Diabetes Mellitus; Arthritis; Foot--Abnormalities; Chronic Obstructive Pulmonary Disease; Obstructive Sleep Apnea; End Stage Renal Disease; Sleep Apnea; Insomnia; Restless Legs Syndrome
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration; Glaucoma; Retinitis Pigmentosa; Vision Disorders; Acute Coronary Syndrome; Heart Failure; Cardiomyopathy, Hypertrophic; Hypotension, Orthostatic; Syncope; Narcolepsy; Dementia; Multiple Sclerosis; Parkinson Disease; Brain Injuries; Spinal Cord Injuries; Stroke; Vertigo; Dizziness; Seizures; Substance-Related Disorders; Diabetes Mellitus, Type 1; Arthritis; Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive; Kidney Failure, Chronic; Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders; Restless Legs Syndrome | interventions — bis(p-chlorophenyl)acetic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Driving Decision Aid (Experimental): Web-based Driving Decision Aid
  Interventions: Behavioral: Driving Decision Aid
- Older Drivers Website (Active Comparator): National Institute on Aging (NIA) Older Drivers website
  Interventions: Behavioral: Older Drivers Website

INTERVENTIONS:
Behavioral: Driving Decision Aid — Healthwise DDA
  Other Names: DDA
  Arms: Driving Decision Aid
Behavioral: Older Drivers Website — National Institute on Aging (NIA) Older Drivers Website
  Arms: Older Drivers Website

SUMMARY:
This Stage II randomized, controlled, longitudinal trial seeks to assess the acceptability, feasibility, and effects of a driving decision aid use among geriatric patients and providers. This multi-site trial will (1) test the driving decision aid (DDA) in improving decision making and quality (knowledge, decision conflict, values concordance and behavior intent); and (2) determine its effects on specific subpopulations of older drivers (stratified for cognitive function, decisional capacity, and attitudinally readiness for a mobility transition). The overarching hypotheses are that the DDA will help older adults make high-quality decisions, which will mitigate the negative psychosocial impacts of driving reduction, and that optimal DDA use will target certain populations and settings.

DETAILED DESCRIPTION:
The investigators will use a multi-site, two-armed randomized controlled trial of older drivers (n=300; ≥70 years) from clinical settings, and one family member each (n=up to 300), with longitudinal follow-up. Study goals are to test how much the DDA improves outcomes and identify who benefits most from the DDA. Evaluation of the DDA's efficacy (Aim 1) and its relative effect in subgroups (Aim 2) corresponds to Stage II in the NIH Stage Model for Behavioral Intervention Development. Findings from Aims 1 & 2 could identify necessary refinements (Stage I) and inform future efficacy, effectiveness or implementation trials.

ELIGIBILITY:
Inclusion Criteria for drivers:

* 70 years or older
* Fluent in English
* At least one medical condition linked in driving cessation
* Drive at least one time per week
* Have a study partner* (*drivers interested in participating in the study without a study partner will be placed on a wait list; they may be contacted as a later date for enrollment once 200 driver-study partner dyads have been enrolled across all sites)
* 5-minute MoCA score greater or equal to 21

Exclusion Criteria for drivers:

* In legal custody or institutionalized
* Significant cognitive impairment as measured by 5-minute Montreal Cognitive Assessment (MoCA)
* Since the last time they had their license renewed, has had at least one major change to health, vision, or hearing that has seriously impaired driving (based on potential participant self-report)
* Feels the Department of Motor Vehicles would have serious concerns about their driving (based on potential participant self-report)

Inclusion Criteria for study partners:

* 18 years or older
* Fluent in English
* Identified by Driver participant to contact for potential participation, i.e., part of a driver-study partner dyad
* 5-minute MoCA score greater or equal to 21

Exclusion Criteria for study partners:

* In legal custody or institutionalized
* Significant cognitive impairment as measured by 5-minute Montreal Cognitive Assessment (MoCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 529 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marian E Betz, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of California, San Diego, La Jolla, California
  - CU Anschutz Medical Center, Aurora, Colorado
  - Indiana University, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansmann KJ, Meuser T, Johnson RL, Peterson RA, Fowler NR, DiGuiseppi C, Han D, Moran R, Omeragic F, Betz ME. Internal Factors that Influence Coping in Older Drivers' Transition to Non-Driving. J Appl Gerontol. 2025 Jul;44(7):1172-1180. doi: 10.1177/07334648241298670. Epub 2024 Dec 3. PMID 39626218
- [Derived] Betz ME, Hill LL, Fowler NR, DiGuiseppi C, Han SD, Johnson RL, Meador L, Omeragic F, Peterson RA, Matlock DD. "Is it time to stop driving?": A randomized clinical trial of an online decision aid for older drivers. J Am Geriatr Soc. 2022 Jul;70(7):1987-1996. doi: 10.1111/jgs.17791. Epub 2022 Apr 20. PMID 35441700
- [Derived] Betz ME, Omeragic F, Meador L, DiGuiseppi CG, Fowler NR, Han SD, Hill L, Johnson RL, Knoepke CE, Matlock DD, Moran R; AUTO Research Team. The Advancing Understanding of Transportation Options (AUTO) study: design and methods of a multi-center study of decision aid for older drivers. Inj Epidemiol. 2021 May 3;8(1):23. doi: 10.1186/s40621-021-00310-4. PMID 33934709

RESULTS

PARTICIPANT FLOW:
Period: Baseline Enrollment (Drivers + SPs)
Arm/Group | Older Drivers Website | Driving Decision Aid
Started | 267 (151 drivers, 116 study partners) | 262 (150 drivers, 112 study partners)
Completed | 267 (151 drivers, 116 study partners) | 262 (150 drivers, 112 study partners)
Not Completed | 0 | 0
Period: 6 Month Follow-up (Drivers Only)
Arm/Group | Older Drivers Website | Driving Decision Aid
Started | 151 (151 drivers (no study partner data collected at this visit)) | 150 (150 drivers (no study partner data collected at this visit))
Completed | 144 (144 drivers (no study partner data collected at this visit)) | 138 (138 drivers (no study partner data collected at this visit))
Not Completed | 7 | 12
Not completed — Missed interview | 3 | 8
Not completed — Withdrawal by Subject | 4 | 4
Period: 12 Month Follow-up (Drivers + SPs)
Arm/Group | Older Drivers Website | Driving Decision Aid
Started | 263 (147 drivers, 116 study partners) | 258 (146 drivers, 112 study partners)
Completed | 242 (139 drivers, 103 study partners) | 224 (131 drivers, 93 study partners)
Not Completed | 21 | 34
Not completed — Missed interview | 9 | 20
Not completed — Death | 1 | 4
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Withdrawn by team | 0 | 2
Period: 18 Month Follow-up (Drivers Only)
Arm/Group | Older Drivers Website | Driving Decision Aid
Started | 143 (143 drivers (no study partner data collected at this visit)) | 143 (143 drivers (no study partner data collected at this visit))
Completed | 129 (129 drivers (no study partner data collected at this visit)) | 123 (123 drivers (no study partner data collected at this visit))
Not Completed | 14 | 20
Not completed — Missed interview | 12 | 14
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Withdrawn by team for health issues/hospitalization | 0 | 1
Period: 24 Month Follow-up (Drivers and SPs)
Arm/Group | Older Drivers Website | Driving Decision Aid
Started | 249 (141 drivers, 108 study partners) | 238 (137 drivers, 101 study partners)
Completed | 218 (125 drivers, 93 study partners) | 211 (125 drivers, 86 study partners)
Not Completed | 31 | 27
Not completed — Missed interview | 22 | 18
Not completed — Death | 2 | 3
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Withdrawn by team due to health issues | 2 | 0

BASELINE CHARACTERISTICS:
Population: Comprised of older adult drivers with 1+ medical condition linked to driving cessation (N = 301) and their family/friends acting as study partners (N = 228)
Groups:
- Total: Total of all reporting groups
Arm/Group | Older Drivers Website | Driving Decision Aid | Total
Number analyzed (Participants) | 267 | 262 | 529
Age, Categorical [Count of Participants; unit: Participants] — Population: N = 1 participant refused to share their age with the study team.
  Participants
    number analyzed (Participants) | 267 | 261 | 528
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 41 | 36 | 77
    >=65 years | 226 | 225 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: N = 1 participant refused to share their age with the study team.
  years
    number analyzed (Participants) | 267 | 261 | 528
    (all) | 71.1 (11.9) | 73.1 (10.6) | 72.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 156 | 304
  Male | 119 | 106 | 225
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 256 | 256 | 512
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 8 | 6 | 14
  White | 246 | 246 | 492
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 267 | 262 | 529
Pre-randomization decision conflict scale (DCS) score) [Mean (Standard Deviation); unit: units on a scale] — Decision conflict scale (DCS) is calculated from 16 items, with each item ranging from 0 (strongly agree) to 4 (strongly disagree). The total score is reported on a 0-100 scale by summing all responses, dividing by 16 and multiplying by 25. Higher scores represent greater levels of uncertainty in decision-making (higher decision conflict = worse outcome), and interventions often aim to reduce decision conflict (lower decision conflict = greater likelihood of implementing a decision = better outcome).
  units on a scale | 18.5 (12.4) | 17.3 (12.5) | 17.9 (12.4)

OUTCOME MEASURES:

1. Primary Outcome: Decisional Conflict Scale (DCS) Scores at Day 0 (Post-intervention)
Description: Decision conflict scale (DCS) is calculated from 16 items, with each item ranging from 0 (strongly agree) to 4 (strongly disagree). The total score is reported on a 0-100 scale by summing all responses, dividing by 16 and multiplying by 25. Higher scores represent greater levels of uncertainty in decision-making (higher decision conflict = worse outcome), and interventions often aim to reduce decision conflict (lower decision conflict = greater likelihood of implementing a decision = better outcome).
Time Frame: Day 0 (Post-intervention)
Population: Drivers post-randomization at baseline visit. Missing N = 8 participants' outcomes (N = 3 control, N = 5 DDA) because they did not respond to one or more questions required to calculate this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 148 | 145
units on a scale | 15.2 (13.3) | 12.3 (12.9)

2. Secondary Outcome: Values Clarity Subscale Score at Day 0 (Post-intervention)
Description: For the values clarity subscale, three decision conflict scale (DCS) items (Likert scale responses from 0 ['strongly agree'] to 4 ['strongly disagree']) are summed, divided by 3 and multiplied by 25; scores range from 0 (extremely clear) to 100 (extremely unclear about personal values); lower scores represent higher values clarity, which is a better outcome. Lower values clarity subscale scores are associated with positive outcomes. The measure will be assessed in drivers immediately following administration of control condition or intervention.
Time Frame: Day 0 (Post-intervention)
Population: Drivers at post-intervention. Missing N = 3 participants' outcomes (N = 2 control, N = 1 DDA) because they did not respond to one or more questions required to calculate this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 149 | 149
units on a scale | 13.8 (15.3) | 12.8 (15.4)

3. Secondary Outcome: Older Adult Driving Safety Knowledge Scores as Assessed by True/False Questions at Day 0 (Post-intervention)
Description: The following true/false questions will be used to examine participants' safe driving knowledge: 1) Older drivers pose a bigger risk to other drivers and pedestrians than younger drivers do; 2) Drivers aged 70 years and older are more likely to be hurt or killed if they are in a crash; 3) There is a milestone age when everyone should stop driving; 4) With age, a person needs more light to see well; 5) Getting lost on familiar roads is a sign that it might be time to stop driving. A higher number of correctly answered questions indicate better outcomes. Knowledge will be defined as the percentage of correct scores of the 5 questions (ranging from 0% [worst outcome] to 100% [best outcome]). The measure will be assessed in drivers immediately following administration of control condition or intervention.
Time Frame: Day 0 (Post-intervention)
Population: Drivers at post-randomization. Missing N = 7 participants' outcomes (N = 5 control, N = 2 DDA) because they did not respond to one or more questions required to calculate this outcome.
Measure: Mean (Standard Deviation); unit: percentage of correct questions
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 146 | 148
percentage of correct questions | 79.9 (18.4) | 88.9 (16.4)

4. Secondary Outcome: Decision Self Efficacy Score at Day 0 (Post-intervention)
Description: The Decision Self-Efficacy Scale will be used to assess decision self efficacy. Scores range from 0 (extremely low self-efficacy; worst outcome) to 100 (extremely high self-efficacy; best outcome). Higher scores indicate better outcomes. The measure will be assessed in drivers immediately following administration of control condition or intervention
Time Frame: Day 0 (Post-intervention)
Population: Drivers post-randomization. Missing N = 3 participants' outcomes (N = 1 control, N = 2 DDA) because they did not respond to one or more questions required to calculate this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 150 | 149
units on a scale | 92.9 (10.3) | 93.2 (9.4)

5. Secondary Outcome: Change in Patient-Reported Outcomes Measurement Information System (PROMIS) 4-item Depression Score
Description: Depression will be measured using the PROMIS Short Form 4-item scale (4a Adult v1.0), with higher PROMIS scores indicating higher depression. PROMIS scores are presented as standardized T-scores (mean=50, standard deviation=10). Lower PROMIS depression scores indicate better outcomes (lower depression).
  Change in depression is calculated as the PROMIS depression score at each time point (6, 12, 18, or 24 months) minus the score at baseline (pre-randomization). Since PROMIS scores at each time point can range from 41.0 to 79.4, change in depression PROMIS scores can range from -38.4 to +38.4. Change-scores > 0 represent increases in depression (poor outcome), and changes <= 0 represent maintained or decreased depression (better outcome).
Time Frame: 6 months, 12 months, 18 months, 24 months
Population: Drivers with any depression change-scores that could be calculated (had to have baseline depression and data at at least one follow-up). Missing N = 12 participants' outcomes (N = 7 control, N = 5 DDA) either of for two reasons: (i) they withdrew from the study between baseline and 6 month follow-up (N = 8 total; N = 4 control, N = 4 DDA) or (ii) they did not respond to one or more questions needed to calculate this outcome at baseline and/or follow-up (N = 4 total; N = 3 control, N = 1 DDA).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 144 | 145
units on a scale
  6 month follow-up (change from baseline): number analyzed (Participants) | 143 | 138
  6 month follow-up (change from baseline) | 0.56 (5.50) | 0.04 (5.42)
  12 month follow-up (change from baseline): number analyzed (Participants) | 138 | 129
  12 month follow-up (change from baseline) | 1.32 (4.58) | 0.26 (5.91)
  18 month follow-up (change from baseline): number analyzed (Participants) | 127 | 123
  18 month follow-up (change from baseline) | 1.46 (5.05) | -1.10 (5.49)
  24 month follow-up (change from baseline): number analyzed (Participants) | 125 | 124
  24 month follow-up (change from baseline) | 1.20 (5.31) | 0.65 (5.81)

6. Secondary Outcome: Change in Ottawa Decision Regret Score
Description: Change in decision regret will be measured by the Ottawa Decision Regret Scale. This validated measure correlates with decision satisfaction and conflict, and overall quality of life. Scored from 0-100, high scores represent higher regret. Lower scores indicate better outcomes.
  Decision regret was measured at 6, 12, 18, and 24 months, so change in decision regret can be calculated from 12 months (vs. 6 months), 18 months (vs. 6 months), and 24 months (vs 6 months). Since decision regret scores range from 0-100, change in decision regret scores range from -100 to + 100, with change-scores <= 0 representing maintenance or decreases in decision regret (positive outcome) and change-scores > 0 representing increased decision regret over time (negative outcome).
Time Frame: 12 months, 18 months, 24 months
Population: Drivers who had 1+ change-score(s) that could be calculated for decision regret (had to have 6 month decision regret and at least one subsequent follow-up). Missing N = 53 participants' outcomes (N = 20 control, N = 33 DDA) because: (i) they withdrew from the study between baseline and 12 months (N = 15; N = 8 control, N = 7 DDA) or (ii) they did not respond question(s) required to calculate this outcome at 6 month and/or subsequent follow-up visits (N = 38 total, N = 12 control, N = 26 DDA).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 131 | 117
units on a scale
  12 month change-score (12 month - 6 month): number analyzed (Participants) | 122 | 111
  12 month change-score (12 month - 6 month) | 3.24 (15.61) | -1.98 (9.57)
  18 month change-score (18 month - 6 month): number analyzed (Participants) | 119 | 105
  18 month change-score (18 month - 6 month) | 2.39 (15.55) | -1.57 (10.59)
  24 month change-score (24 month - 6 month): number analyzed (Participants) | 117 | 107
  24 month change-score (24 month - 6 month) | 1.71 (15.13) | 0.37 (12.47)

7. Secondary Outcome: Change in Life Space Score
Description: Life space is a global measure of mobility and community engagement. The Life-Space Assessment instrument (UAB Study of Aging) is a validated tool assessing recent mobility and function. Composite scores range from 0 (bedbound) to 120 (travel out of town every day without assistance); scores of ≤60 are correlated with lower levels of social participation and higher mortality. Higher scores indicate better outcomes.
  Change in life space can be calculated at 6 months (vs baseline), 12 months (vs baseline), 18 months (vs baseline), and 24 months (vs baseline). Since life space scores range from 0-120, change-scores in life space can range from -120 to +120. Maintained or increased life space (change-scores >= 0) are positive outcomes, and decreased life space (change-scores < 0) are negative outcomes.
Time Frame: 6 months, 12 months, 18 months, 24 months
Population: Drivers who have at least one life space change-score that can be calculated (required to have baseline life space score and data at at least one follow-up). Missing N = 19 participants' outcomes (N = 11 control, N = 8 DDA) because: (i) they withdrew between baseline and 6 month FU (N = 8 total, N = 4 control, N = 4 DDA) or (ii) they did not respond to one or more questions required to calculate this outcome at baseline and/or follow-up visits (N = 11 total, N = 7 control, N = 4 DDA).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 140 | 142
units on a scale
  6 month change-score (6 month - baseline): number analyzed (Participants) | 139 | 134
  6 month change-score (6 month - baseline) | -1.97 (20.77) | -3.10 (20.09)
  12 month change-score (12 month - baseline): number analyzed (Participants) | 131 | 128
  12 month change-score (12 month - baseline) | 2.68 (19.12) | -2.44 (19.15)
  18 month change-score (18 month - baseline): number analyzed (Participants) | 121 | 121
  18 month change-score (18 month - baseline) | 1.93 (21.08) | -0.16 (20.23)
  24 month change-score (24 month - baseline): number analyzed (Participants) | 116 | 119
  24 month change-score (24 month - baseline) | 1.61 (21.95) | -1.91 (19.93)

8. Secondary Outcome: Change in Self-reported Driving Frequency
Description: Self-reported driving frequency will be measured by number of days per week participants drive, with consideration of higher or lower frequency as a positive or negative outcome in the context of participant's intent to drive with lower or higher frequency.
  In the final study survey, this question was reworded, so participants were asked "during the past 6 months, have you reduced the number of days per week you normally drive?" with response options of "yes", "no", "I don't know". Percentage of those who answered "yes" at each time point are reported.
Time Frame: 6 months, 12 months, 18 months, 24 months
Population: Drivers with a driving frequency response at at least one time point (6 months, 12 months, 18 months, and/or 24 months). Missing N = 11 participants' outcomes (N = 6 control, N = 5 DDA) because they (i) withdrew from the study between baseline and 6 month follow-up (N = 8 total, N = 4 control, N = 4 DDA) or (ii) did not respond to this question at any follow-up visits (N = 3 total, N = 2 control, N = 1 DDA).
Measure: Count of Participants; unit: Participants
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 145 | 145
Participants
  Have reduced days/week driving at 6 months: number analyzed (Participants) | 144 | 139
  Have reduced days/week driving at 6 months | 64 | 70
  days/week driving at 12 months: number analyzed (Participants) | 137 | 130
  days/week driving at 12 months | 44 | 45
  days/week driving at 18 months: number analyzed (Participants) | 126 | 121
  days/week driving at 18 months | 32 | 43
  days/week driving at 24 months: number analyzed (Participants) | 121 | 123
  days/week driving at 24 months | 23 | 29

9. Secondary Outcome: Change in Self-reported Situational Driving Avoidance
Description: Driving avoidance in certain situations will be measured by asking participants about their avoidance of riskier driving situations, e.g., nighttime driving, with consideration of avoidance in certain situations as a positive or negative outcome in the context of participant's intent to avoid these situations.
  Avoidance of night driving was worded as: "Using a scale from 1 to 7 where 1 is Not At All Comfortable and 7 is Completely Comfortable, how comfortable do you feel in the following situation?", and the situation presented was "Driving at night?". Higher scores indicate greater comfort with driving at night, and lower scores represent less comfort. Therefore, change-scores can range from -6 to + 6, with change-scores >= 0 indicate maintained or increased comfort with driving at night, and change-scores < 0 indicate reduced comfort in driving at night.
Time Frame: 6 months, 12 months, 18 months, 24 months
Population: Drivers with any situational driving avoidance change-scores that could be calculated (had to have baseline and data at at least one follow-up). Missing N = 11 participants' outcomes (N = 6 control, N = 5 DDA) for two reasons: (i) they withdrew from the study between baseline and 6 month follow-up (N = 8 total; N = 4 control, N = 4 DDA) or (ii) they did not respond to one or more questions needed to calculate this outcome at baseline and/or follow-up (N = 3 total, N = 2 control, N = 1 DDA).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 145 | 145
units on a scale
  6 month change-score (6 month - baseline): number analyzed (Participants) | 144 | 139
  6 month change-score (6 month - baseline) | -0.10 (1.23) | -0.40 (1.15)
  12 month change-score (12 month - baseline): number analyzed (Participants) | 138 | 130
  12 month change-score (12 month - baseline) | -0.38 (1.06) | -0.42 (1.16)
  18 month change-score (18 month - baseline): number analyzed (Participants) | 127 | 122
  18 month change-score (18 month - baseline) | -0.42 (1.19) | -0.53 (1.27)
  24 month change-score (24 month - baseline): number analyzed (Participants) | 125 | 124
  24 month change-score (24 month - baseline) | -0.69 (1.19) | -0.67 (1.16)

10. Secondary Outcome: Occurrence of Driving Cessation
Description: Driving cessation will be measured by asking participants whether they are currently driving; all participants were currently driving at study baseline. Consideration of driving cessation as a positive or negative outcome will be determined in the context of participant's intent to engage in driving cessation. This question was worded as "Do you currently drive?" with response options of "yes" and "no". The numbers reported are those who said "no", which represents driving cessation.
  The wording of this question was added to the study after an early DSMB meeting, so less data are available for it at earlier time points.
Time Frame: 6 months, 12 months, 18 months, 24 months
Population: Drivers with 1 or more time points of data on driving cessation. Missing N = 21 participants' outcomes (N = 8 control, N = 13 DDA) for two reasons: (i) they withdrew from the study between baseline and 6 month (N = 8 total; N = 4 control, N = 4 DDA) or (ii) they did not respond to this question follow-up (N = 13 total, N = 4 control, N = 9 DDA). This question was inadvertently not added to data collection until the 6 month follow-up period, which is why sample sizes were smaller at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 143 | 137
Participants
  6 month: number analyzed (Participants) | 50 | 46
  6 month | 4 | 1
  12 month: number analyzed (Participants) | 105 | 99
  12 month | 2 | 2
  18 month: number analyzed (Participants) | 127 | 123
  18 month | 6 | 5
  24 month: number analyzed (Participants) | 126 | 124
  24 month | 11 | 3

11. Secondary Outcome: Occurrence of Self-reported Crashes
Description: Occurrence of self-reported crashes will be measured by ≥1 crash versus no crashes, where ≥1 crash is a negative outcome.
Time Frame: 6 months, 12 months, 18 months, 24 months
Population: Drivers with 1 or more time points of data on self-reported crashes. Missing N = 10 participants' outcomes (N = 6 control, N = 4 DDA) for two reasons: (i) they withdrew from the study between baseline and 6 month follow-up (N = 8 total; N = 4 control, N = 4 DDA) or (ii) they did not respond to this question follow-up (N = 2 total, N = 2 control, N = 0 DDA).
Measure: Count of Participants; unit: Participants
Arm/Group | Older Drivers Website | Driving Decision Aid
Number analyzed (Participants) | 145 | 146
Participants
  6 month: number analyzed (Participants) | 144 | 139
  6 month | 15 | 9
  12 month: number analyzed (Participants) | 138 | 130
  12 month | 10 | 10
  18 month: number analyzed (Participants) | 127 | 123
  18 month | 10 | 12
  24 month: number analyzed (Participants) | 123 | 124
  24 month | 12 | 13

ADVERSE EVENTS:
Time Frame: 2 years of study from enrollment to follow-up (baseline, 6 month, 12 month, 18 month, 24 month visits)
Description: Possible adverse events: distress during any assessment (driver or study partner), self-reported motor vehicle accident as driver (drivers only) Possible serious adverse events: DMV report of motor vehicle accident (drivers only), inpatient hospitalization (any reason; drivers or study partners); ED visit (any reason; drivers or study partners); death (all causes; driver or study partner)
Arm/Group | Older Drivers Website | Driving Decision Aid
All-Cause Mortality (participants affected / at risk) | 4/267 | 5/262
Serious Adverse Events (participants affected / at risk) | 3/267 | 4/262
Other Adverse Events (participants affected / at risk) | 16/267 | 17/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Older Drivers Website (N=267) | Driving Decision Aid (N=262)
Motor vehicle accident as driver (Injury, poisoning and procedural complications) | 0/151 (0) | 0/150 (0) — DMV report; drivers only
Inpatient hospitalization (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) — Drivers or study partners
Emergency department (ED) visit (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) — Any reason; drivers or study partners
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Older Drivers Website (N=267) | Driving Decision Aid (N=262)
Distress during any assessment (Social circumstances) | 0 (0) | 1 (1) — Driver or study partner
Motor vehicle accident as driver (Injury, poisoning and procedural complications) | 16/151 (16) | 16/150 (18) — Self-reported; drivers only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT04141891/Prot_SAP_000.pdf